CLINICAL TRIAL: NCT02424305
Title: Pharmacokinetics of LEO 43204 Gel in Actinic Keratosis Administered Under Maximal Use Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LP0084-1077
Record Dates: First submitted 2015-04-14; First posted 2015-04-23 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2017-05

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- face: LEO 43204 gel 0.018% (Experimental): 3 days treatment (once daily) on face: LEO 43204 gel 0.018%
  Interventions: Drug: LEO 43204 gel 0.018%
- arm: LEO 43204 gel 0.1% (Experimental): 3 days treatment (once daily) on arm: LEO 43204 gel 0.1%
  Interventions: Drug: LEO 43204 gel 0.1%
- scalp: LEO 43204 gel 0.037% (Experimental): 3 days treatment (once daily) on scalp: LEO 43204 gel 0.037%
  Interventions: Drug: LEO 43204 gel 0.037%

INTERVENTIONS:
Drug: LEO 43204 gel 0.018%
  Arms: face: LEO 43204 gel 0.018%
Drug: LEO 43204 gel 0.1%
  Arms: arm: LEO 43204 gel 0.1%
Drug: LEO 43204 gel 0.037%
  Arms: scalp: LEO 43204 gel 0.037%

SUMMARY:
This is an open-label, uncontrolled, non-randomised multi-centre trial in which 3 parallel groups will be enrolled. The trial includes three active treatment groups. To be eligible for inclusion in this trial, subjects must have at least 15 clinically typical, visible, and discrete actinic keratosis (AKs) on the face, scalp or on the arm within a contiguous area of approximately 250 cm2 of sun-damaged skin.

There will be 3 treatment groups: (1) once daily application of LEO43204 gel 0.018% on the full face for three consecutive days, (2) once daily application of LEO43204 gel 0.1% on the arm on a treatment area of approximately 250 cm2 for three consecutive days and , (3) once daily application of LEO43204 gel 0.037 % on the scalp for three consecutive days.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with 15 or more clinically typical, visible and discrete AKs on either:

   * Full face (corresponding to a treatment area of at least 250 cm2). If subjects have a beard they must shave no later than the day before the first drug application.
   * A contiguous area of approximately 250 cm2 on the arm between wrist and shoulder.
   * Balding scalp (corresponding to a treatment area of approximately 250 cm2). Subjects with sparse hair on the scalp can be enrolled as long as LSR and AK assessments are not compromised.
2. Subject at least 18 years of age.
3. Female subjects of childbearing potential* must be confirmed not pregnant by a negative urine pregnancy test prior to trial treatment.
4. Female subjects of childbearing potential must be willing to use effective contraception at trial entry and until completion.

Exclusion Criteria:

1. Location of the treatment area (full face, full balding scalp, chest, trunk or extremities)

   * within 5 cm of an incompletely healed wound.
   * within 5 cm of a suspected basal cell carcinoma (BCC) or SCC.
2. Previously assigned treatment in this clinical trial or previously participated in a clinical trial in the LEO 43204 programme.
3. Lesions in the treatment area that have: atypical clinical appearance (e.g. cutaneous horns)and/or, recalcitrant disease (e.g., did not respond to cryotherapy on two previous occasions).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of LEO 43204. | Once daily for 3 days
Peak Plasma Concentration (Cmax) of LEO 43204. | Once daily for 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Edward Lain, MD, Principal Investigator — Pflugerville Dermatology Clinical Research
Locations (1):
- Pflugerville Dermatology Clinical Research, Pflugerville, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lain E, Skov T, Hall A. Pharmacokinetics and Safety of Ingenol Disoxate Gel Administered Under Maximum-Use Conditions to Patients With Actinic Keratosis. Clin Drug Investig. 2018 Mar;38(3):249-257. doi: 10.1007/s40261-017-0608-y. PMID 29204958
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en